CLINICAL TRIAL: NCT01428024
Title: An Open, Multi-center Study Evaluating Efficacy, Safety and Injection Technique of Restylane Lip Products for Lip Enhancement and Lip Rejuvenation
Brief Title: Study to Evaluate Efficacy, Safety and Injection Technique of Restylane Lip Volume and Restylane Lip Refresh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 31GE1102
Record Dates: First submitted 2011-08-31; First posted 2011-09-02 (Estimated); Results first posted 2018-10-18 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2013-11

CONDITIONS: Injection Techniques
Keywords: efficacy; safety; Restylane; Lip products; injection techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Restylane Lip Volume (Experimental): Submucosal injections with Restylane Lip Volume. Treatment of up to 1,5 ml product for upper and lower lip, respectively at week 0 and optional at week 2 and 12.
  Interventions: Device: Restylane Lip Volume
- Restylane Lip Refresh (Experimental): Submucosal injections with Restylane Lip Refresh. Treatment of up to 0,5 ml product for upper and lower lip, respectively at week 0 and optional at week 2 and 12.
  Interventions: Device: Restylane Lip Refresh

INTERVENTIONS:
Device: Restylane Lip Volume — Treatment of up to 1,5 ml product for upper and lower lip, respectively at week 0 and optional at week 12.
  Arms: Restylane Lip Volume
Device: Restylane Lip Refresh — Treatment of up to 0,5 ml product for upper and lower lip, respectively at week 0 and optional at week 12.
  Arms: Restylane Lip Refresh

SUMMARY:
The purpose of this study is to demonstrate the efficacy and safety of two new Restylane Lip products, Restylane Lip Volume and Restylane Lip Refresh, and to collect information on the injection technique.

DETAILED DESCRIPTION:
Restylane Lip Volume is intended to be used for lip enhancement and Restylane Lip Refresh is intended to restore hydrobalance and improve skin structure of the lips (referred to as lip rejuvenation in this protocol), respectively. The lidocaine content is designed to reduce the subject's pain during treatment. The objectives of this open, multicenter study are to evaluate efficacy and safety of the products for the studied indications and to collect information on injection techniques used.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 60 years of age.
* Intent to undergo lip augmentation or rejuvenation of both the upper and lower lip.
* Signed informed consent.

Exclusion Criteria:

* Prior surgery or tattoo to the upper or lower lip or lip line.
* Presence of any abnormal lip structure, such as a scar or lump or severe lip asymmetry.
* A history of herpes labialis and an outbreak within four weeks of study entry or with four or more outbreaks in the 12 months prior to study entry.
* Presence of facial hair that may interfere with efficacy evaluations.
* Active skin disease, inflammation or related conditions, such as infection, psoriasis and herpes zoster near or on the area to be treated.
* History of angioedema.
* Previous hypersensitivity to hyaluronic acid or local anesthetics.
* Concomitant anticoagulant therapy and therapy with inhibitors of platelet aggregation within 10 days prior to treatment, or a history of bleeding disorders.
* Cancerous or pre-cancerous lesions in the area to be treated.
* Previous tissue augmenting therapy in the area to be treated with hyaluronic acid (HA) or collagen filler, or laser treatment, during the last 12 months.
* Permanent implant placed in the area to be treated or treatment with non-HA or non-collagen filler in the area to be treated.
* Pregnancy or breast feeding.
* Participation in any other clinical study within 30 days prior to inclusion.
* Other condition preventing the subject to entering the study in the Investigator's opinion e.g. subjects not likely to avoid other facial cosmetic treatments below the level of the lower orbital rim, subjects anticipated to be unreliable or incapable of understanding the study assessment or unrealistic expectations of treatment result.
* Study staff or close relative to study staff (e.g. parents, children, siblings or spouse).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Samuelsson, Med Dr, Principal Investigator — Akademikliniken, Storängsvägen 10, 115 42 Stockholm; Dan Fagrell, Med Dr, Principal Investigator — Göteborgs Plastikirurgiska Center, Fridkullagatan 35 412 65 Göteborg; Pyra Haglund, Med Dr, Principal Investigator — Stureplanskliniken, Lästmakargatan 10, 111 44 Stockholm
Locations (3):
- Sweden (3):
  - Göteborgs Plastikkirurgiska Center, Gothenburg
  - Stureplanskliniken, Stockholm
  - Akademikliniken, Stockholm

RESULTS

PARTICIPANT FLOW:
Groups:
- Restylane LipVolume: Open label
  Restylane Lip Volume : Treatment of up to 1,5 ml product for upper and lower lip, respectively at week 0 and optional at week 12.
- Restylane Lip Refresh: Open label
  Restylane Lip Refresh : Treatment of up to 0,5 ml product for upper and lower lip, respectively at week 0 and optional at week 12.
Period: Overall Study
Arm/Group | Restylane LipVolume | Restylane Lip Refresh
Started | 30 | 30
Completed | 29 | 29
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Restylane LipVolume: Open label
  Restylane Lip Volume : Treatment of up to 1,5 ml product for upper and lower lip, respectively at week 0 and week 12.
- Restylane Lip Refresh: Open label
  Restylane Lip Refresh : Treatment of up to 0,5 ml product for upper and lower lip, respectively at week 0 and week 12.
- Total: Total of all reporting groups
Arm/Group | Restylane LipVolume | Restylane Lip Refresh | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (12.5) | 49.4 (6.4) | 42.8 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: GEIS (Global Esthetic Improvement Scale) Assessed by the Subject at Week 8 After Treatment
Description: To evaluate esthetic change of lips from baseline as judged by the subjects using GEIS. GEIS is a categorical scale with five levels: very much improved, much improved, somewhat improved, no change, worse.
Time Frame: At week 8 - change of lips from baseline
Population: One subject did not perform GEIS evaluation at the 8-week visit and withdrew consent after the visit
Measure: Number (95% Confidence Interval); unit: percentage improved subjects
Groups:
- Restylane Lip Volume: GEIS (Global Esthetic Improvement Scale)subject at 8 weeks (change from baseline).
  Injection with Restylane Lip Volume (a Hyaluronic acid gel)with maximum 1.5 ml for each upper/lower lip.
- Restylane Lip Refresh: GEIS (Global Esthetic Improvement Scale)subject at 8 weeks (change from baseline).
  Injection with Restylane Lip Refresh (a Hyaluronic acid gel)with maximum 0.5 ml for each upper/lower lip.
Arm/Group | Restylane Lip Volume | Restylane Lip Refresh
Number analyzed (Participants) | 29 | 30
percentage improved subjects | 86.2 [68.3 to 96.1] | 86.7 [69.3 to 96.2]

2. Secondary Outcome: GEIS (Global Esthetic Improvement Scale) Assessed by the Subject at Week 36 After Treatment
Description: To evaluate esthetic change of lips from baseline as judged by the subjects using GEIS at week 36. GEIS is a categorical scale with five levels: very much improved, much improved, somewhat improved, no change, worse.
Time Frame: week 36 - change from baseline
Population: Restylane Lip Volume: One subject withdrew consent after the 8-week visit and thus did not perform the GEIS evaluation at 36 weeks.
  Restylane Lip Refresh: Two subjects did not perform the GEIS evaluation at 36 weeks.
Measure: Number (95% Confidence Interval); unit: percentage improved subjects
Groups:
- Restylane Lip Volume: GEIS (Global Esthetic Improvement Scale) subject at 36 weeks (change from baseline).
  Injection with Restylane Lip Volume (a Hyaluronic acid gel) with maximum 1.5 ml for each upper/lower lip.
- Restylane Lip Refresh: GEIS (Global Esthetic Improvement Scale) subject at 36 weeks (change from baseline).
  Injection with Restylane Lip Refresh (a Hyaluronic acid gel) with maximum 0.5 ml for each upper/lower lip.
Arm/Group | Restylane Lip Volume | Restylane Lip Refresh
Number analyzed (Participants) | 29 | 28
percentage improved subjects | 93.1 [77.2 to 99.2] | 78.6 [59.0 to 91.7]

3. Secondary Outcome: GEIS (Global Esthetic Improvement Scale) Assessed by the Treating Investigator at Week 36 After Treatment
Description: To evaluate esthetic change of lips from baseline as judged by the treating investigator using GEIS at week 36. GEIS is a categorical scale with five levels: very much improved, much improved, somewhat improved, no change.
Time Frame: week 36 - change from baseline
Measure: Number (95% Confidence Interval); unit: percentage improved subjects
Groups:
- Restylane LipVolume: GEIS (Global Esthetic Improvement Scale)by treating investigator at 36 weeks (change from baseline).
  Injection with Restylane Lip Volume (a Hyaluronic acid gel)with maximum 1.5 ml for each upper/lower lip.
- Restylane Lip Refresh: GEIS (Global Esthetic Improvement Scale)by treating investigator at 36 weeks (change from baseline).
  Injection with Restylane Lip Refresh (a Hyaluronic acid gel)with maximum 0.5 ml for each upper/lower lip.
Arm/Group | Restylane LipVolume | Restylane Lip Refresh
Number analyzed (Participants) | 29 | 29
percentage improved subjects | 82.8 [64.2 to 94.2] | 82.8 [64.2 to 94.2]

4. Secondary Outcome: GEIS (Global Esthetic Improvement Scale) Assessed by the Independent Evaluator at Week 36 After Treatment
Description: To evaluate esthetic change of lips from baseline as judged by the independent evaluator using GEIS at week 2, 4, 12, 26 and 36. GEIS is a categorical scale with five levels: very much improved, much improved, somewhat improved, no change, worse.
Time Frame: week 36 - change from baseline
Measure: Number (95% Confidence Interval); unit: percentage improved subjects
Groups:
- Restylane LipVolume: GEIS (Global Esthetic Improvement Scale)independent evaluator at 36 weeks (change from baseline).
  Injection with Restylane Lip Volume (a Hyaluronic acid gel)with maximum 1.5 ml for each upper/lower lip.
- Restylane Lip Refresh: GEIS (Global Esthetic Improvement Scale)independent evaluator at 36 weeks (change from baseline).
  Injection with Restylane Lip Refresh (a Hyaluronic acid gel)with maximum 0.5 ml for each upper/lower lip.
Arm/Group | Restylane LipVolume | Restylane Lip Refresh
Number analyzed (Participants) | 29 | 29
percentage improved subjects | 86.2 [68.3 to 96.1] | 86.2 [68.3 to 96.1]

5. Secondary Outcome: MLFS (Medicis Lip Fullness Scale) at Week 8
Description: To evaluate the efficacy in terms of Medicis Lip Fullness Scale (MLFS) score by live assessment performed separately by the treating and the independent investigators in the Restylane Lip Volume group. The scale has five levels: Very thin, thin, median, full, very full. Treatment success is defined as at least one grade increase.
Time Frame: week 8 - change from baseline
Measure: Number (95% Confidence Interval); unit: percentage improved subjects
Groups:
- Restylane LipVolume: MLFS (Medicis Lip Fullness Scale)score by live assessment performed separately by the treating and the independent investigators at 8 weeks (change from baseline).
  Injection with Restylane Lip Volume (a Hyaluronic acid gel)with maximum 1.5 ml for each upper/lower lip.
Arm/Group | Restylane LipVolume
Number analyzed (Participants) | 30
percentage improved subjects | 50.0 [31.3 to 68.7]

6. Secondary Outcome: Subject Satisfaction Questionnaire
Description: To evaluate subjects satisfaction in terms of a subject satisfaction questionnaire at week 8 after treatment.
  The subject satisfaction questionnaire consists of questions regarding the looks, appearance, disomfort, and satisfaction regarding the treatment of the lips.
  The question that will be referred to is: How satisfied are you today with (the look of) your lips ?
Time Frame: Week 8
Measure: Number; unit: percentage satisfied subjects
Groups:
- Restylane LipVolume: Subject satisfaction questionnaire at 8 weeks. Injection of Restylane Lip Volume (a Hyaluronic acid gel) maximum dosage of 1.5 ml per upper/lower lip.
- Restylane Lip Refresh: Subject satisfaction questionnaire at 8 weeks. Injection of Restylane Lip Refresh (a Hyaluronic acid gel) maximum dosage of 0.5 ml per upper/lower lip.
Arm/Group | Restylane LipVolume | Restylane Lip Refresh
Number analyzed (Participants) | 29 | 30
percentage satisfied subjects | 93 | 87

7. Secondary Outcome: Subject Diary for 14 Days After Initial Treatment
Description: To evaluate the acute safety profile (bruising, itching, pain, redness, swelling and tenderness) in terms of a 14-day subject diary after initial treatment.
  Subjects still reporting one or more of the symptoms; bruising, itching, pain, redness, swelling and tenderness in the diary at day 14.
Time Frame: 2 weeks after initial treatment
Measure: Number; unit: participants
Groups:
- Restylane Lip Volume: Open label
  Restylane Lip Volume : Treatment of up to 1,5 ml product for upper and lower lip, respectively at week 0 and optional at week 12.
Arm/Group | Restylane Lip Volume | Restylane Lip Refresh
Number analyzed (Participants) | 30 | 30
participants | 2 | 6

ADVERSE EVENTS:
Arm/Group | Restylane LipVolume | Restylane Lip Refresh
Serious Adverse Events (participants affected / at risk) | 3/30 | 0/30
Other Adverse Events (participants affected / at risk) | 16/30 | 21/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restylane LipVolume (N=30) | Restylane Lip Refresh (N=30)
Knee joint injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Viral encephalitis (Infections and infestations) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Worsening of benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restylane LipVolume (N=30) | Restylane Lip Refresh (N=30)
Lip dry (Gastrointestinal disorders) | 2 (4) | 1 (1)
Implant site haematoma (General disorders) | 5 (9) | 9 (12)
Implant site mass (General disorders) | 7 (10) | 7 (8)
Implant site pain (General disorders) | 2 (3) | 0 (0)
Implant site swelling (General disorders) | 2 (4) | 7 (10)
Injection site pain (General disorders) | 3 (4) | 1 (1)
oral herpes (Infections and infestations) | 1 (1) | 2 (2)
Blood blister (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Implant site erythema (General disorders) | 0 (0) | 2 (2)
Implant site haemorrhage (General disorders) | 1 (1) | 3 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less